CLINICAL TRIAL: NCT02139059
Title: Staged Ureteroscopy After Initial Urinary Drainage Versus Direct Ureteroscopy in the Treatment of Pediatric Obstructive Calcular Anuria
Brief Title: Delayed or Direct Ureteroscopy in the Treatment of Pediatric Calcular Anuria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohammed said elsheemy, Associte professor of urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61179
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Acute Renal Failure; Anuria; Obstructive Uropathy; Ureteric Stones
Keywords: anuria; children; ureteroscopy; initial urinary drainage; ureteric stones
MeSH Terms: conditions — Acute Kidney Injury; Anuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- initial urinary drainage (Active Comparator): initial urinary drainage to stabilize renal functions before ureteroscopy
  Interventions: Procedure: initial urinary drainage
- direct ureteroscopy (Active Comparator): direct ureteroscopy without initial urinary drainage
  Interventions: Procedure: direct ureteroscopy

INTERVENTIONS:
Procedure: initial urinary drainage — initial urinary drainage is done using nephrostomy or double J stent to stabilize renal functions. this is followed several days later by definitive ureteroscopy.
  Arms: initial urinary drainage
Procedure: direct ureteroscopy — direct ureteroscopy is done without initial urinary drainage and before return to normal chemistry. this is followed follow-up of renal functions for several days before treatment of the contralateral side.
  Arms: direct ureteroscopy

SUMMARY:
To compare staged ureteroscopy following initial urinary drainage versus direct ureteroscopy without initial urinary drainage in the treatment of obstructive calcular anuria with acute renal failure in children.

DETAILED DESCRIPTION:
To compare staged ureteroscopy following initial urinary drainage and stabilization of renal functions using percutaneous nephrostomy or double J stent versus direct ureteroscopy without initial urinary drainage in the treatment of obstructive calcular anuria with acute renal failure due to ureteric calculi in children.

ELIGIBILITY:
Inclusion Criteria:

* children ≤12 years old presenting with Obstructive Anuria and Acute Renal Failure due to bilateral ureteric stones suitable for ureteroscopy.

Exclusion Criteria:

* Fever, pyonephrosis or sepsis.
* unstable patients are stabilized first by dialysis.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Return to normal creatinine | 1 week
  period for return to normal creatinine in both groups
stone free status | 1 week
  success in removal of ureteric stones using ureteroscopy
operative and early post operative complications | 1 week
  Hematuria, Extravasation (perforation), mucosal complications, stone migration, failure of ureteric access, fever

SECONDARY OUTCOMES:
ureteric stricture | 6 months
  occurrence of ureteric stricture as a delayed complication
period to reach stone free status bilaterally | 6 months
  period to reach stone free status bilaterally after the treatment of the contralateral side
number of times of exposure to general anesthesia | 6 months
  number of times of exposure to general anesthesia during successive interventions to clear stones bilaterally

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S ElSheemy, A professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt